CLINICAL TRIAL: NCT01474928
Title: Asthma and Health Literacy in Newcomer Communities in the Greater Vancouver Area (GVA): A Population-based Qualitative Study
Brief Title: Asthma and Health Literacy in Newcomer Communities in the Greater Vancouver Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government); Ministry of Health, British Columbia (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mark Fitzgerald, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H08-02861; 187972 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Asthma; Community-based participatory research; Educational intervention; Ethno-cultural community; Video recording; Patient education handout
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 2: community video group (Experimental): In each community intervention group two subject viewed the patient role played community video
  Interventions: Behavioral: patient role played community video; Behavioral: Community video group
- Group three: both videos group (Experimental): In each community intervention group three subject viewed two videos (the patient role played community and physician-led knowledge videos)
  Interventions: Behavioral: both videos group
- Group four: pamphlet group (Active Comparator): In each community intervention group four subject read an educational pamphlet only - act as active comparator group
  Interventions: Behavioral: Pamphlet group
- Group one: knowledge video group (Experimental): In each community intervention group one subject viewed the physician-led knowledge video
  Interventions: Behavioral: physician-led knowledge video; Behavioral: knowledge video

INTERVENTIONS:
Behavioral: patient role played community video — Group two viewed the patient role played community video
  Arms: Group 2: community video group
Behavioral: both videos group — Group three viewed both the knowledge and community videos
  Arms: Group three: both videos group
Behavioral: Pamphlet group — Group four read an educational pamphlet only
  Arms: Group four: pamphlet group
Behavioral: physician-led knowledge video — Group one viewed a physician-led knowledge video
  Arms: Group one: knowledge video group
Behavioral: Community video group — Group two viewed the patient role played community video
  Arms: Group 2: community video group
Behavioral: knowledge video — Group one viewed a physician-led knowledge video
  Arms: Group one: knowledge video group

SUMMARY:
In this study, the investigators aim to develop and test the effectiveness of culturally appropriate asthma videos and other educational materials based on knowledge from this study and the investigators' previous studies. By culturally appropriate materials the investigators mean to develop health information (in the format of video and written materials) in the community own language and applied the most appealing cultural beliefs and practices in the Chinese and Punjabi communities. The investigators also aim to recommend a practical framework and to develop a measure of asthma knowledge and health literacy among immigrants from the Punjabi and Chinese communities in BC. The investigators' definition of health literacy in this study is the capability of a person to navigate and access to asthma-related information, as well as to understand, evaluate, and communicate the obtained information to improve his/her health status. The investigators' hypothesis is that audio-visual based asthma information in a subject's native language would improve a patient's knowledge and self-management of asthma in comparison to printed information.

DETAILED DESCRIPTION:
There is compelling evidence indicating that newcomers to Canada with limited English proficiency and low health literacy are facing systemic, linguistic and cultural barriers in accessing health information and treatment services pertaining to Asthma. The intent of this study is to develop and test the effectiveness of culturally appropriate asthma videos and other educational materials based on knowledge from this study and the investigators' previous elicitation studies, to recommend a practical framework and to develop a measure of asthma knowledge and health literacy among immigrants from the Punjabi and Chinese communities in the Greater Vancouver Area.

The objectives of the proposed research are: "1." to assess the knowledge, attitudes, beliefs, and practices related to asthma and relevant issues in selected individuals within the target communities; "2." to investigate access and utilization patterns of asthma-related services among participant communities; "3." to assess the effectiveness of culturally competent and participatory developed videos and written educational materials on individuals' knowledge and health literacy skills related to asthma; "4." to examine relationships between health literacy, culture, language and access to and utilization of asthma services among targeted newcomer individuals; "5." to build research capacity and community-university-service provider alliances, and contribute to the development of an integrated research-service agenda on newcomers' asthma self-management among target communities; and "6." to disseminate information to decision makers and knowledge-users , so the results of this study can be efficiently used in developing relevant services that meet newcomers' needs. The proposed research will use quantitative and qualitative methods including a full participatory approach that builds on the investigators' previous work with vulnerable ethno-cultural communities in BC.

The implementation of the project will include the following phases:

"1." Conduct environmental scan and needs assessment study (literature review and interviews); "2" Develop video clips, written materials, and relevant measurement tools; "3" Apply the video clips and written materials to test their effectiveness among individuals from the target communities in terms of asthma self-management; "4" Conduct quantitative and qualitative data analysis; and "5" Disseminate the findings to larger audiences, key-informants, knowledge users and policy makers across BC. This research will make theoretical, methodological and applied research contributions. It will establish strong community - academic connections for the development of the proposed framework. Community participation will be applied throughout the development of this study and educational materials, enhancing the potential of acquiring new knowledge about cultural and traditional practices of the sample population.

The investigators' approach will allow health care workers and policy makers to design appropriate health promotion initiatives targeted to diverse newcomer groups in relation to asthma. The investigators foresee findings that provide not only better ways to measure health literacy pertaining to asthma in the investigators' target groups, but that will also help develop materials and measures that can be applied to diverse cultural populations in BC and the rest of Canada. The investigators expect that the participatory approach used in this study will contribute to capacity building, improving newcomers' ability to access and use relevant asthma information (in terms of prevention, control and management) and to transfer and share the information learned with other members of the target communities. The proposed community consultation will also help the investigators to identify culturally appropriate communication mode(s) to deliver health promotion messages and determine practical adult learning approaches applicable to diverse communities in Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosed mild to moderate asthma according to CTS criteria
2. Asthmatics from Chinese and Punjabi communities in the Greater Vancouver Area (GVA), BC
3. Age greater than 21 years
4. Immigrated to Canada in the last 10 yrs
5. Patients who are able to give informed consent and are willing to participate in the study

Exclusion Criteria:

1. Age less than 21 years
2. Other immigrants than Punjabi and Chinese
3. Immigrated before 1998
4. Patients who do not want to sign the consent form

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-08; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
medication adherence | on year
  Patients' understanding of physicians' instructions on how to follow their treatment regimen and regular use of inhalers were measured

SECONDARY OUTCOMES:
Patients' beliefs, perceptions, and attitudes toward asthma self-management | 6 months
  The investigators aimed to explore both broad and specific issues and concerns about asthma and its management of the patients from the target communities
Educational materials and measurement tools development | 3 months
  The investigators involved end-users (i.e. asthma patients, their family members, and community key-informants) in developing linguistically and culturally appropriate education materials (e.g., video clips and pictorial pamphlets) and measurement tools, and conducted community events and forums.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J FitzGerald, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Centre for Clinical Epidemiology and Evaluation, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia

REFERENCES:
- [Result] Poureslami I, Rootman I, Doyle-Waters MM, Nimmon L, Fitzgerald JM. Health literacy, language, and ethnicity-related factors in newcomer asthma patients to Canada: a qualitative study. J Immigr Minor Health. 2011 Apr;13(2):315-22. doi: 10.1007/s10903-010-9405-x. PMID 20938742
- [Result] Poureslami I, Shum J, Nimmon L, FitzGerald JM. Evaluating effect of culturally-specific educational interventions on asthma subjects' inhaler use technique and their understanding of physician instructions. Respiratory care, 2016
- [Derived] Poureslami I, Tregobov N, Shum J, McMillan A, Akhtar A, Kassay S, Starnes K, Mahjoob M, FitzGerald JM. A conceptual model of functional health literacy to improve chronic airway disease outcomes. BMC Public Health. 2021 Jan 30;21(1):252. doi: 10.1186/s12889-021-10313-x. PMID 33516200
- [Derived] Poureslami I, Shum J, Nimmon L, FitzGerald JM. Culturally Specific Evaluation of Inhaler Techniques in Asthma. Respir Care. 2016 Dec;61(12):1588-1596. doi: 10.4187/respcare.04853. Epub 2016 Nov 8. PMID 27827331
- [Derived] Poureslami I, Nimmon L, Doyle-Waters M, Rootman I, Schulzer M, Kuramoto L, FitzGerald JM. Effectiveness of educational interventions on asthma self-management in Punjabi and Chinese asthma patients: a randomized controlled trial. J Asthma. 2012 Jun;49(5):542-51. doi: 10.3109/02770903.2012.682125. PMID 22715910
- See also: British Columbia Centre for Lung Health — http://www.centreforlunghealth.ca
- See also: The Lung Centre at University of British Columbia — http://www.thelungcentre.ca/